CLINICAL TRIAL: NCT01617395
Title: Integrating Genetic and Environmental Risk Scores Into an Algorithm to Predict Multiple Sclerosis Susceptibility
Brief Title: Relating Genetic and Environmental Risk Scores to Multiple Sclerosis Susceptibility
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120122; 12-N-0122
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-11-24

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Magnetic Resonance Imaging (MRI); Natural History
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GEMS cohort: Individuals at risk for developing MS
- Healthy volunteer cohort: healthy volunteers, ages 18-50, who do not have a known first-degree relative with MS
- MS patient cohort: MS patients whose first-degree relatives are enrolled in this study

SUMMARY:
Background:

- Research shows that both genes and the environment influence a person s risk for getting multiple sclerosis (MS). However, it is not possible to accurately predict who will develop MS. Researchers want to study people with MS and their family members. They have developed a Genetic and Environmental Risk Score for MS. This score combines information from a person's medical history and genes. It also includes environmental factors that may be related to developing MS. This study will test this risk score to see if it can help predict who will develop MS.

Objectives:

- To evaluate a score for genetic and environmental risk factors that may help predict whether a person will develop MS.

Eligibility:

* Individuals at least 18 years of age who have MS.
* Individuals between 18 to 50 years of age who are the parent, brother, sister, or child of a person with MS.

Design:

* People with MS will allow researchers to look at their personal and medical data. These data will have been collected in other MS-related studies.
* Relatives of people with MS will fill out a questionnaire and give blood and saliva samples. They will fill out the questionnaire again one year later.
* Some relatives will have additional optional testing. These tests will include a physical exam and imaging studies. There may also be other tests. These tests may be repeated every 1 to 5 years for 20 years.

DETAILED DESCRIPTION:
Objective. The overall objective of this study is to investigate the genetic, immune, and neuroimaging profiles that may increase a person s risk of developing multiple sclerosis (MS) in order to identify and validate predictive biomarkers in populations at risk for this disorder.

Study population. There will be three study populations:

1. Individuals at risk for developing MS As part of the Genes and Environment in Multiple Sclerosis (GEMS) study, we plan to recruit up to 1000 first-degree relatives of MS patients. GEMS is a study aiming to recruit 5000 individuals that is being led by our collaborators at Columbia University Medical Center. For the purposes of this study, a first-degree relative may be a parent, sibling, or child between 18 and 50 years of age but must not carry a diagnosis of MS. The first-degree relative must have the ability to provide consent and be willing to participate in the study. Two potentially overlapping subsets of these individuals will undergo detailed testing at the NIH:

   1. The cross-sectional subcohort will consist of up to 150 participants with combined genetic and environmental risk scores (GERS), defined in the protocol, in the highest and lowest 20 percent of the entire study population. Selected participants may be invited for follow-up studies based on data obtained at baseline if symptoms develop.
   2. The NINDS longitudinal subcohort will consist of up to 10 participants, ages 18 to 40,who express willingness to be followed for 20 years at the NIH, whose GERS falls in the top 20 percent of the entire study population, and who have a first-degree relative with MS who is participatipate
2. MS patients - We plan to recruit up to 1000 MS patients whose first-degree relatives are enrolled this study. These participants either: (A) will be evaluated under other Neuroimmunology Branch Clinic protocols and will not undergo separate evaluation under this protocol; or (B) will send us medical records confirming their MS diagnosis via mail/fax/secure email, without the requirement to participate in another NIH protocol. The purpose of including this cohort in the current study is to allow access to their clinical, biological, and imaging data for comparison with first-degree relatives, if available, and to confirm that existing GEMS participants have a first-degree relative diagnosed with MS.
3. Healthy volunteers - We plan to recruit up to 80 healthy volunteers, ages 18-50, who do not have a known first-degree relative with MS. The purpose of including this cohort in the current study is to allow quantification of the degree and extent of abnormalities, including abnormalities of the blood-brain barrier, in individuals at risk for developing MS. Without imaging data obtained from healthy volunteers, there is no way to determine whether subtle clinical and neuroimaging findings in the at-risk cohort are truly abnormal, or to correctly threshold and quantify the observed abnormalities.

Design. This is a prospective cohort natural-history study. All GEMS participants will complete the following study procedures, which can be performed offsite: informed consent; study questionnaire; saliva sample; and blood draw. The questionnaire will be repeated 1 year after enrollment.

There will two additional substudies conducted at NIH: a cross-sectional substudy and a longitudinal substudy. Participants in these substudies will be evaluated with clinical, radiological, and laboratory procedures. Participants in the cross-sectional cohort will undergo evaluation at the NIH at a single time point (with optional longitudinal follow up), whereas participants in the longitudinal cohort will undergo evaluation at the NIH for 20 years. There will be an interim analysis 5 years after the 50th participant is recruited to the longitudinal cohort, and the study of this cohort may be terminated if we have not observed the development of MS-related radiological or laboratory abnormalities in any of the participants. Participants with MS will provide informed consent to allow access to their own research data, but the data themselves will be (or will have already been) collected under other Neuroimmunology Clinic clinical protocols.

NIH is a unique site within the overall GEMS study, for the following reasons: (1) It is the only site at which imaging is being performed, as part of the cross-sectional and longitudinal substudies; (2) GEMS participants seen at NIH may undergo additional procedures that are not part of the overall GEMS study; (3) Data from participants in the NIH substudy will be directly linked to data from their own relatives with MS.

Outcome measures. For participants in the overall GEMS study, the primary outcome measure is the GERS itself, as most participants in this cohort will not undergo further testing. For participants in the cross-sectional cohort, which consists of individuals at highest and lowest risk for MS, the primary outcome measure is the presence or absence of lesions on T2-weighted brain MRI that meet the 2010 MRI criteria for dissemination in space - a finding that, in this population, may well be related to MS. For participants in the longitudinal cohort, the study endpoint is a clinical diagnosis of MS according to the same 2010 criteria. Secondary outcome measures include: (1) The age at which participants develop MS-related abnormalities on brain imaging studies, abnormalities on laboratory testing, and clinical symptoms and signs; (2) The time lag between defined exposures (for example, infectious mononucleosis) and the appearance of MS-related radiological, laboratory, and clinical abnormalities; (3) The time lag between the appearance of asymptomatic radiological and laboratory abnormalities and the onset of clinical symptoms; and (4) Additional exploratory clinical, imaging, and biological data in the crosssectional that may suggest subclinical MS disease activity.

ELIGIBILITY:
* INCLUSION CRITERIA:

GEMS cohort (target n equals 1000)

* First-degree relative (parent, sibling, or child) of a self-reported MS patient.
* Age 18-50, inclusive, at the time of enrollment into the overall GEMS study.
* Willingness to be contacted regarding additional follow-up procedures.
* Cross-sectional subcohort (target n equal 150):

  * Referred by Columbia University Medical Center as having a genetic and environmental risk score (GERS), defined in Section 4.1.1, in the top or bottom 20% of the overall GEMS study.
* NINDS Longitudinal subcohort (target n equal 100):

  * Ages 18-40, inclusive.
  * Referred by Columbia University Medical Center as having a GERS in the top 20% of the overall GEMS study.
  * Willing to undergo additional study procedures at the NIH for up to 20 years, with planned follow-up every year for participants between ages 18 and 25, every 2 years for participants between ages 26 and 30, and every 5 years for participants between ages 31 and 40.
  * Relative enrolled in NIH study with confirmation of MS diagnosis.

MS patient cohort (target n=1000):

* MS patients (NIH)

  * Co-enrolled in another Neuroimmunology Clinic natural history protocol.
  * Diagnosis confirmed at NIH.
  * Age 18 or older.
* MS patient (non-NIH)

  * First-degree relative (parent, sibling, or child) of an existing GEMS participant.
  * Able and willing to send medical records associated with their MS diagnosis to NIH.
* Healthy volunteer cohort (target n=80)

  * Age 18-50, inclusive.
  * No known first-degree relative (parent, sibling, or child) with MS.
* All cohorts

  * Able to give informed consent.

EXCLUSION CRITERIA:

GEMS cohort

-Diagnosis of MS.

Cross-sectional and NINDS longitudinal subcohorts

* Contraindications to MRI scanning.
* Diagnosis of another central nervous system disease disease (CNS neoplasm, known cerebrovascular disease, known CNS degenerative diseases, or known CNS inflammatory diseases) at the time enrollment into the study.
* MS cohort (both)

  --None
* Healthy volunteer cohort

  * Diagnosis of MS or another central nervous system (CNS neoplasm, cerebrovascular disease CNS degenerative diseases, or CNS inflammatory diseases) or a systemic disease that would interfere with the aims of this study.
  * Contraindications to MRI scanning.

Eligible NIH employees and staff may participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2012-08-15 (Actual)

PRIMARY OUTCOMES:
presence or absence of lesions on T2-weighted brain MRI | ongoing
  For participants in the cross-sectional cohort, which consists of individuals at highest and lowest risk for MS, the primary outcome measure is the presence or absence of lesions on T2-weighted brain MRI that meet the 2010 MRI criteria for dissemination in space.
GERS | ongoing
  For participants in the overall GEMS study, the primary outcome measure is the GERS itself, as most participants in this cohort will not undergo further testing.

SECONDARY OUTCOMES:
The time lag between the appearance of asymptomatic radiological and laboratory abnormalities and the onset of clinical symptoms; | ongoing
  The time lag between the appearance of asymptomatic radiological and laboratory abnormalities and the onset of clinical symptoms;
The time lag between defined exposures | ongoing
  time lag between defined exposures (for example, infectious mononucleosis) and the appearance of MS-related radiological, laboratory, and clinical abnormalities
exploratory clinical, imaging, biological data in the cross sectional | ongoing
  exploratory clinical, imaging, and biological data in the cross sectional that may suggest subclinical MS disease activity
development of MS-like abnormalities on brain imaging studies, abnormalities on laboratory testing, and clinical symptoms and signs. | ongoing
  The age at which participants develop MS-related abnormalities on brain imaging studies, abnormalities on laboratory testing, and clinical symptoms and signs;

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is not a clinical trial

REFERENCES:
- [Background] Ascherio A, Munger KL, Lennette ET, Spiegelman D, Hernan MA, Olek MJ, Hankinson SE, Hunter DJ. Epstein-Barr virus antibodies and risk of multiple sclerosis: a prospective study. JAMA. 2001 Dec 26;286(24):3083-8. doi: 10.1001/jama.286.24.3083. PMID 11754673
- [Background] Balcer LJ. Clinical practice. Optic neuritis. N Engl J Med. 2006 Mar 23;354(12):1273-80. doi: 10.1056/NEJMcp053247. No abstract available. PMID 16554529
- [Background] Chiappa KH. Use of evoked potentials for diagnosis of multiple sclerosis. Neurol Clin. 1988 Nov;6(4):861-80. PMID 3070342
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-N-0122.html